CLINICAL TRIAL: NCT02881892
Title: Interleukin-6, Procalcitonin and Vascular Endothelial Growth Factor in Plasma and Dialysate Correlate With Peritoneal Solute Transport and Dialysis Adequacy in CAPD Patients
Brief Title: Iplasma IL6, Procalcitonin and VEGF and Dialysate Level in CAPD Patients
Status: Completed | Type: Observational
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Other Study IDs: 041/57
Record Dates: First submitted 2016-08-18; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Kidney Disease
Keywords: CAPD; Peritoneal solute transport rate; Dialysis adequacy
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Procalcitonin; Vascular Endothelial Growth Factor A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Measure plasma and dialysate level of IL-6, procalcitonin and VEGF — correlation between plasma levels, dialysate appearance rate of VEGF, inflammatory cytokines (IL- 6, procalcitonin) and PSTR, dialysis adequacy in CAPD patients.

SUMMARY:
The aim of study was to evaluated the correlation between plasma levels, dialysate appearance rate of VEGF, inflammatory cytokines (IL- 6, procalcitonin) and PSTR, dialysis adequacy in CAPD patients.

DETAILED DESCRIPTION:
This cross -sectional study measured IL-6, procalcitonin and VEGF level in plasma and overnight effluent. PSTR of small solutes was evaluated by standard peritoneal equilibration test (standard PET). Weekly Kt/V and creatinine clearance (CCr ) were evaluated in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Stable CAPD patients without previous history of peritonitis

Exclusion Criteria:

* HIV
* Other infections, tuberculosis or on immunosuppressive drugs,
* Autoimmune disease,
* Cancer
* Diagnosis of permanent ultrafiltration failure .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CAPD patients age more than 18 years
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
plasma level of VEGF, IL-6 and procalcitonin with the PSTR and dialysis adequacy in CAPD patients | 2 years
  measure in pg/ml

SECONDARY OUTCOMES:
Cytokines in diabetic and non-diabetic group | 2 years
  All cytokines in plasma and blood

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvniach, M.D., Principal Investigator — Department of Medicine,Vajira Hospital,Navamindradhiraj University
Locations (1):
- Renal Unit, BMA Medical College and Vajira Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh KH, Jung JY, Yoon MO, Song A, Lee H, Ro H, Hwang YH, Kim DK, Margetts P, Ahn C. Intra-peritoneal interleukin-6 system is a potent determinant of the baseline peritoneal solute transport in incident peritoneal dialysis patients. Nephrol Dial Transplant. 2010 May;25(5):1639-46. doi: 10.1093/ndt/gfp670. Epub 2010 Jan 8. PMID 20061317
- [Background] Alscher DM, Mettang T. Procalcitonin in peritoneal dialysis--a useful marker of inflammation? Perit Dial Int. 2005 Sep-Oct;25(5):441-4. No abstract available. PMID 16178476
- [Background] Herget-Rosenthal S, Klein T, Marggraf G, Hirsch T, Jakob HG, Philipp T, Kribben A. Modulation and source of procalcitonin in reduced renal function and renal replacement therapy. Scand J Immunol. 2005 Feb;61(2):180-6. doi: 10.1111/j.0300-9475.2005.01545.x. PMID 15683455
- [Background] Guz G, Colak B, Hizel K, Reis KA, Erten Y, Bali M, Sindel S. Procalcitonin and conventional markers of inflammation in peritoneal dialysis patients and peritonitis. Perit Dial Int. 2006 Mar-Apr;26(2):240-8. PMID 16623432
- [Result] Pecoits-Filho R, Araujo MR, Lindholm B, Stenvinkel P, Abensur H, Romao JE Jr, Marcondes M, De Oliveira AH, Noronha IL. Plasma and dialysate IL-6 and VEGF concentrations are associated with high peritoneal solute transport rate. Nephrol Dial Transplant. 2002 Aug;17(8):1480-6. doi: 10.1093/ndt/17.8.1480. PMID 12147798